CLINICAL TRIAL: NCT01517841
Title: Barriers to Selection and Initiation of Peritoneal Dialysis in the United States
Brief Title: Barriers to Peritoneal Dialysis Selection
Status: Completed | Type: Observational
Sponsor: MetroHealth Medical Center (Other)
Responsible Party: Principal Investigator, Ash Sehgal, Professor, MetroHealth Medical Center
Other Study IDs: IRB11-00542
Record Dates: First submitted 2012-01-20; First posted 2012-01-25 (Estimated); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Chronic Kidney Disease
Keywords: peritoneal dialysis; modality choice; kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic kidney disease: Patients with chronic kidney disease (20% or less kidney function remaining. Patients with end stage renal disease who are currently receiving dialysis.

SUMMARY:
The purpose of this study is to understand what prevents chronic kidney disease patients from making a timely decision about dialysis modality options. This understanding will allow us to develop and implement interventions to assist patients in this turning point so that they can make the right decision for them in a timely enough manner so that each patient can start dialysis in the safest and best way for them. 200 later stage chronic kidney disease patients (20% or less of kidney function remaining) will be asked to participate in the study with the goal of having 150 patients participate in the study.

Hypotheses:

1. 50 % of patients will have made a modality decision when interviewed and patients in the action stage of behavior will be more likely to make a modality selection than patients in earlier stages of behavior change. Barriers to modality selection will act at several levels including patient, provider and health system level and will vary by behavioral stage of change
2. 10-15% of patients might choose home dialysis. Knowledge, self efficacy in terms of CKD, education, and income will likely be barriers to home dialysis choice.

ELIGIBILITY:
Inclusion Criteria:

* All patients of age greater than or equal to 18 years at MHMC who are late stage CKD

Exclusion Criteria:

* Patients who have acute renal failure and then recover renal function to levels of eGFR (estimated glomerular filtration rate) 20 mL/min/1.73m2 and in whom the nephrologist feels will not progress to ESRD in 2 years
* Patients who are not candidates for peritoneal dialysis
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients with late stage CKD and ESRD patients who are cared for by nephrologists at MetroHealth Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Barriers to making a dialysis modality decision | 1 year
  Determine the proportion of patients that made a dialysis modality decision and determine the barriers to being able to make a decision. Determine the proportion of patients choosing home dialysis and barriers associated with choice of home dialysis therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Suma Prakash, MD, Principal Investigator — MetroHealth Medical Center
Locations (1):
- MetroHealth Medical Center- Center for Reducing Health Disparities, Cleveland, Ohio, United States